CLINICAL TRIAL: NCT07196085
Title: Neural Mechanisms and Efficacy of Imagery Rescripting for Fear of Failure: A Randomized Controlled Neuroimaging Trial
Brief Title: Neural Mechanisms and Efficacy of Imagery Rescripting for Fear of Failure
Acronym: JM2019b
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Sciences and Humanities, Warsaw (Other)
Responsible Party: Principal Investigator, Jaroslaw Michalowski, Professor, University of Social Sciences and Humanities, Warsaw
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SONATA_BIS_JM2019b
Record Dates: First submitted 2025-09-18; First posted 2025-09-29 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Fear of Failure
Keywords: Fear of failure; Imagery Rescripting; Skin Conductance Level; fMRI

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imagery Rescripting (Experimental): Four ImRs sessions over 2 weeks, targeting autobiographical criticism memory. Therapist-guided rescripting involved modifying the "hotspot" scene (critical interaction) with protective interventions addressing unmet needs.
  Interventions: Behavioral: Imagery Rescripting
- Sham Neutral Imagery (Active Comparator): Four neutral imagery sessions over 2 weeks. Participants imagined neutral interpersonal interactions matched in structure and duration to ImRs but with rescription of neutral instead of criticism memories.
  Interventions: Behavioral: Sham Neutral Imagery

INTERVENTIONS:
Behavioral: Imagery Rescripting — Four ImRs sessions over 2 weeks, targeting autobiographical criticism memory. Therapist-guided rescripting involved modifying the "hotspot" scene (critical interaction) with protective interventions addressing unmet needs.
  Arms: Imagery Rescripting
Behavioral: Sham Neutral Imagery — Four neutral imagery sessions over 2 weeks. Participants imagined neutral interpersonal interactions matched in structure and duration to ImRs but with rescription of neutral instead of criticism memories.
  Arms: Sham Neutral Imagery

SUMMARY:
This randomized controlled trial investigates the neural and psychophysiological mechanisms of Imagery Rescripting (ImRs) in individuals with high fear of failure. Participants (N=81, aged 21-34) were randomized to ImRs or an active control condition. The intervention targeted autobiographical memories of parental criticism across four sessions delivered within two weeks. Neuroimaging (fMRI), skin conductance, and self-report measures were assessed pre- and post-intervention (accordindly, TP1, TP5), with follow-ups at 3 and 6 months (accordingly, TP6, TP7). The primary aim was to examine whether ImRs reduces neural and subjective reactivity to autobiographical criticism memories and whether prediction error or memory reconsolidation disruption underlie therapeutic effects.

DETAILED DESCRIPTION:
Fear of failure is a common psychological problem often associated with parental criticism and maladaptive perfectionism. Imagery Rescripting (ImRs) is a therapeutic technique derived from schema therapy that aims to modify distressing autobiographical memories by introducing corrective experiences in imagination. While ImRs has shown efficacy in anxiety and personality disorders, its underlying neural mechanisms remain insufficiently understood.

This randomized controlled neuroimaging trial investigated the effects of ImRs on autobiographical memories of criticism in young adults with high levels of fear of failure. The study specifically examined whether therapeutic change is driven by disruption of memory reconsolidation or by prediction error mechanisms, both of which have been proposed as key pathways for updating maladaptive memories.

Participants (N=81, aged 21-34) meeting inclusion criteria for high fear of failure (Performance Failure Appraisal Inventory ≥ 108) were randomized in a 2:1 ratio to either an ImRs intervention group or an active control group. Exclusion criteria included psychiatric disorders (e.g., PTSD, major depression), active pharmacotherapy, history of childhood abuse, and contraindications to MRI.

All participants underwent two fMRI sessions (pre- and post-intervention), four intervention sessions within a two-week period, and follow-up assessments at 3 and 6 months. During fMRI, participants listened to personalized autobiographical scenarios: five involving parental criticism and five neutral ones. In the ImRs group, the criticism scenario was modified by introducing an imagined therapist figure who interrupted the critical interaction, addressed the child's needs, and suggested alternative positive outcomes. In the control group, participants engaged in a structurally similar neutral imagery task without therapeutic modification.

Primary outcomes included changes in neural activation (BOLD fMRI) in fear-related brain regions (amygdala, thalamus, insula, ventromedial prefrontal cortex) when processing criticism versus neutral memories. Secondary outcomes included functional connectivity between prefrontal and subcortical regions, subjective ratings of arousal and emotions during scenarios, and questionnaire-based measures of fear of failure, perfectionism, and failure-related schemas. An exploratory outcome examined activation of the caudate nucleus during rescripting as a neural correlate of prediction error.

The trial aimed to clarify whether ImRs reduces emotional reactivity at neural and subjective levels, and whether therapeutic effects are mediated reconsolidation-related neural changes or by prediction error. By combining personalized autobiographical stimuli, fMRI, psychophysiological measures, and longitudinal follow-up, the study provides novel insights into the mechanisms of memory-focused psychotherapy in individuals at risk of maladaptive perfectionism and fear of failure.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18-35
* high fear of failure
* not currently undergoing psychotherapy or psychopharmacotherapy
* no severe punitive experiences in the past

Exclusion Criteria:

* current severe affective disorders
* current severe anxiety
* current severe personality disorders
* active suicidality
* psychosis
* substance abuse

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
BOLD fMRI activation to autobiographical criticism scenarios | Pre-treatment (TP1) and 2-weeks post-treatment (TP5).
  Blood-oxygen-level dependent (BOLD) signal in fear-related regions (amygdala, thalamus, insula, vmPFC) during listening to criticism vs. neutral autobiographical scenarios. Contrasts analyzed for anticipation (ANT), hotspot (HOT), and combined phases.
Performance Failure Appraisal Inventory (PFAI) | Screening, pre-treatment (TP1), 2-weeks post-treatment (TP5), 3- & 6-month follow-up (TP6, TP7)
  The Performance Failure Appraisal Inventory was used to assess fear of failure. It is a 35-item questionnaire that measures the strength of subjective beliefs about the consequences of failure. The PFAI has five subscales: fear of experiencing shame and embarrassment; fear of devaluing one's self-esteem; fear of having an uncertain future; fear of important others losing interest, and fear of upsetting important others, with scores ranging 35-175. Higher scores indicate higher level of fear of failure.
Functional connectivity (fMRI) | Pre-treatment (TP1) and 2-weeks post-treatment (TP5)
  Psychophysiological interaction (PPI) and ROI-to-ROI connectivity between vmPFC/dlPFC and fear-related subcortical regions (amygdala, insula, thalamus, hippocampus, PCC, ACC, precuneus) during criticism vs. neutral autobiographical scenarios.
Subjective ratings at the end of all sessions | Pre-treatment (TP1), 2-weeks post-treatment (TP5), 3- & 6-month follow-up (TP6, TP7)
  Subjective ratings at the end of all sessions - participants were asked to evaluate each fragment of the presented scenarios according to several measures: immersion, focus, emotions (happiness, sadness, guilt, fear, anger, disgust) on a 9-point Likert scale (very low-very high), and valence (very negative-very positive), scores ranging 1-9 for each factor.
Failure-related Schemas (FA-YSQ) | Pre-treatment (TP1), 2-weeks post-treatment (TP5), 3- & 6-month follow-up (TP6, TP7).
  Failure-related subscale of the Young Schema Questionnaire (YSQ). Higher scores indicate stronger maladaptive beliefs about failure. Scores ranges from 0 to 54.
Frost Multidimensional Perfectionism Scale (FROST) | Pre-treatment (TP1), 2-weeks post-treatment (TP5), 3- & 6-month follow-up (TP6, TP7).
  35-item questionnaire assessing perfectionism dimensions: Personal Standards, Organization, Concern Over Mistakes, Doubts About Actions, Parental Expectations, and Parental Criticism. Scores range 35-175. Higher scores indicate higher level of perfectionism.
SCL recordings | Screening, pre-treatment (TP1), 2-weeks post-treatment (TP5), 3- & 6-month follow-up (TP6, TP7)
  Skin conductance level (SCL) was collected during the audio-guided scenarios' imagery at pre-treatment, treatment, post-treatment, and follow-up sessions. SCL was acquired using Biopack MP160 EDA-MRI system, with a sampling frequency of 2000Hz. The signal was resampled into 1000Hz, then smoothed with median (100 samples), and filtered with a high-passed 1Hz filter. We calculated normalized change in SCL with equation 100#(SCLStim-SCLbaseline/SCLbaseline), where SCLStim is the mean signal value during the stimulus and SCLbaseline is an SCL reaction during the baseline preceding the first part in each scenario (Sugimine et al., 2020). Our primary outcome was SCL during the imagery of different scenarios, separated for anticipation and hotspot parts.

SECONDARY OUTCOMES:
Working Alliance Inventory (WAI, short form) | 6-month follow-up (TP7).
  Assesses therapeutic alliance between participant and therapist across three domains: bond, goals, and tasks. Rated after final intervention. Score ranges from 0 to 60, with higher scores indicating higher working alliance.
Beck Depression Inventory | Screening, 6-month follow-up
  Beck Depression Inventory second edition (BDI-II) is a self-report scale using 21 items regarding the presence and strength of depression symptoms, with scores ranging 0-63. Higher levels of BDI indicate higher level of depressive symtpoms.
Yale-Brown Obsessive-Compulsive | Screening, 6-month follow-up
  Yale-Brown Obsessive-Compulsive self-report severity scale Y-BOCS-SR a 10-item, self-report questionnaire created to evaluate OCD severity, scores ranging 0-40 (higher scores indicate higher level of OCD symptoms).
M.I.N.I. Mini International Neuropsychiatric Interview | Screening
  M.I.N.I. Mini International Neuropsychiatric Interview is a short structured interview for DSM IV and ICD 10 disorders, used to assess mental disorders: major depressive disorder, dysthymic disorder, suicidality, mania, panic disorder, agoraphobia, social phobia, specific phobia, obsessive-compulsive disorder, post-traumatic stress disorder, alcohol dependence/abuse, drug dependence/abuse, antisocial personality disorder. Based on positive answers to questions clinician diagnose adequate disorders.
Social Anxiety Disorder Scale (DSM) | Screening, 6-month follow-up
  Self-report dimensional scale for Social Anxiety Disorder based on DSM-5 criteria. The scale consists of 10 items measuring frequency of symptoms experienced in the last 7 days. Each item is rated on a 4-point Likert scale (0 = never, 4 = all the time). Scores range 0-40, with higher scores indicating greater symptom severity.
Panic Disorder Scale (DSM) | Screening, 6-month Follow-up (TP7)
  10-item self-rating questionnaire based on DSM-5 criteria for Panic Disorder. The scale assesses symptom frequency over the past 7 days using a 4-point Likert scale (0-4), with total scores ranging from 0 to 40.
Generalized Anxiety Disorder Scale | Screening, 6-month Follow-up (TP7)
  A dimensional measure for Generalized Anxiety Disorder based on DSM-5, comprising 10 items. Participants indicate how frequently they experienced each symptom during the past 7 days. Scoring is on a 4-point Likert scale from 0 (never) to 4 (all the time), with total scores ranging 0-40.
Post-Traumatic Stress Symptoms Scale (DSM) | Screening, 6-month Follow-up (TP7)
  Self-report scale assessing PTSD symptoms as defined by DSM-5 criteria. The instrument includes 10 items evaluating symptom frequency over the previous 7 days on a 0-4 Likert scale. Total scores range from 0 to 40, with higher scores indicating higher symptoms severity.
Structured Clinical Interview for DSM-5 (SCID-5-PD) | Screening
  Structured Clinical Interview for DSM-5 SCID-5-PD is a semistructured clinical interview that evaluates DSM-5 personality disorders under three clusters of A, B, and C, and other specific personality disorders. Based on positive answers to questions clinician diagnose adequate personality disorders.
Drug Abuse Screen Test | Screening
  Drug Abuse Screen Test DAST 10 is a self-reported questionnaire to detect drug use disorders, scores ranging 0-10. Higher scores indicates higher level of drug usage.

CONTACTS AND LOCATIONS:
Overall Officials: Jarosław M. Michałowski, PHD, Principal Investigator — Poznań Laboratory of Affective Neuroscience, Institute of Psychology, SWPS
Locations (1):
- Poznań Laboratory of Affective Neuroscience, Institute of Psychology, SWPS University, Warsaw, Poland, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data from this study, including questionnaire responses, psychophysiological recordings (skin conductance), and neuroimaging data (NIfTI format), as well as analytic code, have already been deposited in the institutional repository (SWPS University Science Cloud). These data are available for secondary analyses by other researchers.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The de-identified dataset was made publicly available 22 September 2025 and will remain accessible indefinitely.
Access Criteria: The data used for analysis (in the form of questionnaires, psychophysiological, and neuroimaging measures) are openly available in the SWPS University repository under a Creative Commons license (CC BY-SA). Access to some raw data (e.g., unprocessed MRI files or full physiological recordings) may be granted upon reasonable request and with permission of the study's principal investigator.
URL: https://share.swps.edu.pl/entities/dataset/5a766acb-f567-43c2-8e65-14db3d4346f7

REFERENCES:
- [Background] Conroy, D. E., Willow, J. P., & Metzler, J. N. (2002). Multidimensional fear of failure measurement: The performance failure appraisal inventory. Journal of applied sport psychology, 14(2), 76-90.
- [Background] Agren T, Engman J, Frick A, Bjorkstrand J, Larsson EM, Furmark T, Fredrikson M. Disruption of reconsolidation erases a fear memory trace in the human amygdala. Science. 2012 Sep 21;337(6101):1550-2. doi: 10.1126/science.1223006. PMID 22997340
- [Background] Arntz A, Weertman A. Treatment of childhood memories: theory and practice. Behav Res Ther. 1999 Aug;37(8):715-40. doi: 10.1016/s0005-7967(98)00173-9. PMID 10452174
- [Background] Morina N, Lancee J, Arntz A. Imagery rescripting as a clinical intervention for aversive memories: A meta-analysis. J Behav Ther Exp Psychiatry. 2017 Jun;55:6-15. doi: 10.1016/j.jbtep.2016.11.003. Epub 2016 Nov 9. PMID 27855298
- [Background] Schiller D, Kanen JW, LeDoux JE, Monfils MH, Phelps EA. Extinction during reconsolidation of threat memory diminishes prefrontal cortex involvement. Proc Natl Acad Sci U S A. 2013 Dec 10;110(50):20040-5. doi: 10.1073/pnas.1320322110. Epub 2013 Nov 25. PMID 24277809
- [Background] Siegesleitner M, Strohm M, Wittekind CE, Ehring T, Kunze AE. Improving imagery rescripting treatments: Comparing an active versus passive approach. J Behav Ther Exp Psychiatry. 2020 Dec;69:101578. doi: 10.1016/j.jbtep.2020.101578. Epub 2020 Jun 9. PMID 32569854
- [Background] Sugimine S, Saito S, Takazawa T. Normalized skin conductance level could differentiate physical pain stimuli from other sympathetic stimuli. Sci Rep. 2020 Jul 2;10(1):10950. doi: 10.1038/s41598-020-67936-0. PMID 32616939
- [Background] Craske MG, Kircanski K, Epstein A, Wittchen HU, Pine DS, Lewis-Fernandez R, Hinton D; DSM V Anxiety; OC Spectrum; Posttraumatic and Dissociative Disorder Work Group. Panic disorder: a review of DSM-IV panic disorder and proposals for DSM-V. Depress Anxiety. 2010 Feb;27(2):93-112. doi: 10.1002/da.20654. PMID 20099270